CLINICAL TRIAL: NCT02485340
Title: The Effect of Sumatriptan and Placebo on Isosorbide-5-mononitrate Induced Headache. Development of a Pragmatic Migraine Model
Brief Title: The Effect of Sumatriptan and Placebo on Isosorbide-5-mononitrate Induced Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Emma Katrine Hansen, Medical doctor, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-6-2014-071
Record Dates: First submitted 2015-06-04; First posted 2015-06-30 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — isosorbide-5-mononitrate; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sumatriptan (Active Comparator): headache is induced with 5-ISMN. This headache is treated double-blinded with 1 tablet of sumatriptan 50 mg
  Interventions: Drug: 5-ISMN (isosorbide-5-mononitrate); Drug: Sumatriptan
- Placebo (Placebo Comparator): headache is induced with 5-ISMN. This headache is treated double-blinded with 1 tablet of placebo (the tablet is similar to the active tablet)
  Interventions: Drug: 5-ISMN (isosorbide-5-mononitrate); Drug: Placebo

INTERVENTIONS:
Drug: 5-ISMN (isosorbide-5-mononitrate) — 5-ISMN is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Other Names: Imdur
Drug: Sumatriptan — 5-ISMN is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Other Names: Imigran
  Arms: Sumatriptan
Drug: Placebo — 5-ISMN is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Arms: Placebo

SUMMARY:
To develop a pragmatic migraine model the investigators will induce headache in healthy volunteers and in patients with migraine without aura with a long lasting Nitrogen Oxide (NO) donor. If the headache responds to sumatriptan, the model can be used to test new drug candidates.

DETAILED DESCRIPTION:
There remains a great need for more effective anti-migraine drugs with fewer side effects. Human experimental models are valuable in early phase development of new anti-migraine drugs but useful models have not yet been developed. The investigators' group has shown that Isosorbide-5-mononitrate (5-ISMN), a long lasting NO-donor, induce headache/migraine in both healthy volunteers and in patients with migraine without aura (MO). To validate this model, the headache must respond to specific migraine treatment with sumatriptan.

Hypothesis: 5-ISMN induces a migraine-like headache in both healthy subjects and in MO-patients and induced headache responds to a specific anti migraine drug; sumatriptan.

Aim: Developing a pragmatic and valid model for the testing of new anti-migraine drugs

ELIGIBILITY:
Inclusion Criteria:

Healthy:

* healthy subjects of both sexes
* age 18-70 years
* weight 50-90 kg.
* Females were requested to use effective contraception.

Migraine patients:

* Migraine patients who meet International headache society (IHS) criteria for migraine with or without aura of both sexes
* 18-70 years
* 45-95 kg.

Exclusion Criteria:

Healthy:

* Any type of headache (except episodic tension-type headache < 1 day per week)
* Serious somatic or psychiatric disease
* Pregnancy
* Intake of daily medication (except oral contraceptives).

Migraine patients:

* Any other type of headache then migraine without aura (except episodic tension-type headache < 1 day per week)
* Serious somatic or psychiatric disease
* Pregnancy, and intake of daily medication (except oral contraceptives).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Median headache score 0 hours after sumatriptan/placebo | 0 hours
Median headache score 2 hours after sumatriptan/placebo | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Emma Katrine Hansen, Doctor, Principal Investigator — Danish Headache Center
Locations (1):
- Emma Katrine Hansen, Copenhagen, Glostrup, Denmark